CLINICAL TRIAL: NCT00307281
Title: Emphysema Research Registry; Screening Study and Genetic Testing
Brief Title: Emphysema Research Registry and Biosample Repository
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Frank C Sciurba, Director, Emphysema/COPD Research Center, University of Pittsburgh
Other Study IDs: STUDY19120059; ERC Registry (Registry Identifier: Emphysema COPD Research Registry and Biosample Reposiory)
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Emphysema; Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The DNA studies that will be done as a part of this study will be restricted to/used for studies of genetics associated with COPD. Optional Alpha-1 Antitrypsin swab testing will also be performed on COPD subjects.
  Specimens will assigned a study ID#
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Registry: 10 pack year tobacco smoking history required, current or former smokers accepted.

SUMMARY:
The Comprehensive Lung Center (CLC) at the University of Pittsburgh Medical Center (UPMC Health System) provides patients with any type of breathing or lung disorder a full range of diagnostic and therapeutic services. The Emphysema/COPD Research Center (ECRC) is a specialty clinic, within this center, that attempts to advance the understanding of emphysema and to evaluate new therapies for patients with emphysema. The Emphysema Research Registry will enable pulmonary research physicians to: 1) gather information and create a research registry of people who have been diagnosed with emphysema; 2) utilize this research registry with the purpose of conducting research that attempts to advance the understanding of emphysema and to evaluate new therapies; and, 3) use the research registry to identify potential candidates for future research programs. These aims will be achieved by the collection of DNA (genetic material)for analysis and storage in addition to pulmonary function tests and other medical information.

DETAILED DESCRIPTION:
The Emphysema/COPD Research Center will enroll up to 3000 subjects at the University of Pittsburgh. The experimental procedures that will be conducted as a part of the Emphysema Research Registry include gathering basic personal information (e.g., name, address, phone number, etc.), asking basic screening questions (which may involve the examination of past, current, and future medical records with an authorized release and the collection of personally identifiable medical record information), completing two breathing questionnaires, performing screening lung function tests to determine breathing capacity and blood oxygen levels, to have blood drawn, to complete a measurement of leg muscle strength, and to have a measurement of body fat.

The breathing questionnaires are known as the St. George's Respiratory Questionnaire (SGRQ), the Medical Research Council Dyspnea Questionnaire (MRCDQ) and COPD assessment Test (CAT). These are paper and pencil questionnaires that inquire about respiratory symptoms, quality of life, and shortness of breath.

Breathing tests are routine clinical tests that measure lung function; spirometry (measures the ability to move air in and out of the lungs), lung volumes (measures the amount of air trapped in the lungs), diffusing capacity (measures how well lungs transfer oxygen to blood), forced oscillometry testing (measures respiratory resistance), and pulse oximetry (measures blood oxygen levels). In addition, subjects will be asked to inhale two puffs of albuterol, which is an inhaled medicine (bronchodilator) that may open up breathing passages, and to repeat some of the breathing tests.

The initial blood work will consist of two samples. The first sample will examine routine tests such as blood chemistries (such as sodium and potassium), hemoglobin, blood count, and blood sugar. The second sample will involve DNA testing. The DNA in your cells is what determines your genetic makeup. The DNA studies that will be done for this Research Registry will be restricted to studies of genetics associated with COPD. The total amount of blood drawn will be 5 tablespoons or less. A separate consent form, Consent 2, addresses this second blood draw in detail. In addition to the initial blood draw, the participant will be asked to contact the center when they are experiencing a COPD exacerbation (increased cough, change in sputum, shortness of breath, etc.). At that time, the participant will be asked to either come to the clinic or allow a study coordinator to go to them and obtain an additional sample of blood. The total amount of this sample will be less than 2 tablespoons. Biologic samples (serum plasma) will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e. name, social security number, birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. Biological samples may (or will or will not) be given to investigators outside of UPMC or may be utilized in future studies.

Leg muscle strength will be measured using an isokinetic dynamometer (MERAC, Universal, Cedar Rapids, IA) in all subjects. Strength will be measured as peak angular force (Newton-m) generated at an angular velocity of 60º/sec during three maximal continuous repetitions. Subjects will be provided standardized instructions and perform practice maneuvers to ensure smooth torque curves.

Body fat testing, also known as Fat Free Mass (FFM) testing, will be measured using a single frequency bioelectrical impedance method in the supine position, as the mean of two measurements (one on each side of the body), using equipment previously used by the Emphysema Research Center (BIA 101/s RJL-Systems, Detroit, MI). The FFM index will be calculated by dividing FFM by height in meters2 as an accurate measure of muscle mass.

All study procedures including Informed Consent, breathing questionnaires, breathing tests, blood work, leg muscle strength testing, and body fat testing will be conducted at the Emphysema/COPD Research Center, located in Suite 1211, Kaufmann Building. The informed consent usually takes 30 minutes, the Patient Data Form will require 5 minutes to fill out, the two breathing questionnaires will take 15 minutes, the screening lung function tests usually take less than 1 hour, the blood work will take 15 minutes, the leg muscle strength testing will take 10 minutes, and the body fat testing will take 5 minutes.

The information from each subject will be entered into the Emphysema Research Registry. The information will be held here until a research protocol is developed or an outside investigator approaches Dr. Frank C. Sciurba. The information gathered (basic personal information, basic screening questions, breathing questionnaires, screening lung function tests, blood work, leg muscle strength, and body fat) will be updated periodically, based on investigator need.

ELIGIBILITY:
Inclusion Criteria:

* Patients would be required to have COPD based on at least one of the following: clinical history, pulmonary function results, or radiographic results.

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current and former smokers with a 10 pack year tobacco history.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2000-08 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
To gather information and create a research registry of people who have been diagnosed with emphysema and a control cohort of research participants without lung diseases, | Indefinite
  This research registry will allow us to to advance the understanding of emphysema and to evaluate new therapies for patients with emphysema.

SECONDARY OUTCOMES:
To continue communications with past, present, and future research participants. | Indefinite
  To utilize this research registry with the purpose to learn more about the pathogenesis of emphysema and the efficacy of new therapies, and to provide a mechanism for improving the quality of treatment for emphysema and advance the field.

CONTACTS AND LOCATIONS:
Overall Officials: Frank C. Sciurba, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Emphysema/COPD Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided